CLINICAL TRIAL: NCT07045545
Title: A Multicenter Randomized Controlled Trial Comparing Platelet-Rich Fibrin and Ventral Dartos Flap as Intermediate Layers in Tabularized Incised Plate (TIP) Urethroplasty for Distal Hypospadias With Mild Penile Curvature
Acronym: PRF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Medical Center, Uzbekistan (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Zafar Abdullaev, Head of Pediatric urology department at National Childrens' Medical Center, Tashkent, Uzbekistan, National Children's Medical Center, Uzbekistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0620251
Record Dates: First submitted 2025-06-10; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: PRF; Hypospadias; Distal Hypospadias; Hypospadias Repair; Fistula Stenosis; Cosmetic Outcomes; Functional Outcomes; Tubularized Incised Plate
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: PRF applied over neourethra; (Experimental): * In patients randomized to the PRF group (Group A), autologous platelet-rich fibrin will be prepared intraoperatively using the following standardized protocol:
  * Approximately 10 minutes before completion of urethroplasty, a 5-10 mL peripheral blood sample to be drawn from the cephalic vein under sterile conditions. The blood to be immediately transferred into a plain sterile glass tube without anticoagulants or additives. Centrifugation to be performed at 3000 rpm (approximately 400×g) for 10 minutes using a bench-top centrifuge.
  * Following centrifugation, three distinct layers were formed:
    1. Acellular plasma (top)
    2. Platelet-rich fibrin clot (middle)
    3. Red blood cells (bottom)
  * The PRF clot to be carefully extracted using sterile forceps , and residual red blood cells were gently separated to ensure a clean PRF membrane. The PRF clot will then gently compressed between saline-soaked sterile gauze to form a pliable membrane suitable for surgical application.
  Interventions: Procedure: - Group A: Platelet-rich fibrin membrane prepared intraoperatively and applied over neourethra
- Group B: Ventral dartos flap rotated over neourethra (Active Comparator): Participants in this arm will undergo hypospadias repair with the application of a ventral dartos fascia flap. The procedure involves elevating a vascularized flap of ventral dartos fascia from the penile shaft, rotating it over the neourethra to provide additional tissue coverage and promote healing. This flap helps in reducing the risk of fistula formation and enhances vascular support to the neourethra. The surgical steps include dissecting the dartos fascia carefully, rotating it over the neourethral reconstruction, and securing it in place, followed by standard postoperative care and follow-up.
  Interventions: Procedure: Group B: Ventral dartos flap rotated over neourethra

INTERVENTIONS:
Procedure: - Group A: Platelet-rich fibrin membrane prepared intraoperatively and applied over neourethra — In this arm, a platelet-rich fibrin membrane will be prepared intraoperatively from the patient's blood using centrifugation. The prepared PRF membrane will then be applied directly over the neourethra following urethroplasty to promote healing and tissue regeneration.
  Arms: Group A: PRF applied over neourethra;
Procedure: Group B: Ventral dartos flap rotated over neourethra — Participants in this arm will undergo hypospadias repair with the application of a ventral dartos fascia flap. The procedure involves elevating a vascularized flap of ventral dartos fascia from the penile shaft, rotating it over the neourethra to provide additional tissue coverage and promote healing. This flap helps in reducing the risk of fistula formation and enhances vascular support to the neourethra. The surgical steps include dissecting the dartos fascia carefully, rotating it over the neourethral reconstruction, and securing it in place, followed by standard postoperative care and follow-up.
  Arms: Group B: Ventral dartos flap rotated over neourethra

SUMMARY:
Distal hypospadias is the most common form of hypospadias. The Tubularized Incised Plate (TIP) repair is the standard surgical technique for this condition; however, complications such as fistula formation and meatal stenosis remain concerns. These complications are often influenced by the choice of intermediate tissue layer used to reinforce the neourethra. The traditional ventral dartos flap is effective but can be technically challenging and may result in a bulky tissue layer.

Platelet-rich fibrin (PRF) is an autologous, growth factor-rich biological material that has shown promise in tissue regeneration and healing. It is easy to prepare intraoperatively and may serve as a biological reinforcement to reduce postoperative complications.

This study aims to provide high-quality evidence comparing the effectiveness of PRF versus the ventral dartos flap in patients with distal hypospadias, specifically those with Grade 1 urethral defects and minimal penile curvature, using a stratified study population to ensure balanced groups.

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the incidence of urethrocutaneous fistula at a minimum of 6 months postoperatively between two intermediate layers used in hypospadias repair: platelet-rich fibrin (PRF) membrane and ventral dartos flap. The study will also evaluate secondary outcomes, including rates of meatal stenosis, urethral stricture, other postoperative complications, and cosmetic outcomes assessed by standardized photographs and blinded expert scoring.

Study Design and Setting:

This prospective, multicenter, single-blinded randomized controlled trial will be conducted at centers in Tashkent, Uzbekistan, and Jakarta, Indonesia. A total of 140 patients (70 per group) will be enrolled, with randomization stratified by urethral plate score and center to ensure balanced groups.

Participants:

Children aged 6 months to 5 years with primary distal hypospadias (Grade 1, Abbas classification) or redo distal hypospadias (Grade 1, Abbas classification), with penile curvature less than 30° after degloving (measured as per Abbas, 2022), will be included. Exclusion criteria include previous hypospadias surgery, proximal hypospadias, penile curvature ≥30°, or syndromic anomalies/coagulopathies.

Interventions:

Participants will undergo tubularized incised plate (TIP) or glanuloplasty TIP (GTIP) urethroplasty performed by experienced pediatric urologists using standardized techniques.

Group A: Application of autologous platelet-rich fibrin membrane over the neourethra. PRF will be prepared intraoperatively by drawing 10 mL of peripheral blood, centrifuging at 3000 rpm for 10 minutes, extracting the PRF clot, compressing it into a membrane, and securing it over the neourethra with absorbable sutures.

Group B: Rotation of a ventral dartos flap over the neourethra.

Intraoperative PRF Preparation:

Blood will be collected into sterile glass tubes without anticoagulants, centrifuged immediately, and the PRF membrane prepared as described. The membrane will be placed over the neourethra before glans closure, secured laterally, and the skin closure completed in standard fashion.

Stratification:

Participants will be stratified based on urethral plate characteristics using a validated scoring system before randomization to ensure anatomical balance.

Follow-Up:

Patients will be assessed at 1, 3, and 6 months postoperatively for complications (fistula, stenosis, etc.), neomeatus function, and cosmetic appearance. Digital photographs will be evaluated by two blinded pediatric urologists, and cosmetic outcomes will be scored using the HOSE system.

Data Management and Analysis:

All data will be anonymized and stored securely. Statistical analysis will be performed using SPSS v22, applying appropriate tests for categorical and continuous variables, with multivariate regression if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Primary and complex distal hypospadias (Grade 1, Abbas classification)
2. Penile curvature <30° after degloving (Methodology of curvature measurement: Abbas T. O. (2022).
3. Children aged 6 months to 5 years

Exclusion Criteria:

1. Previous hypospadias surgery
2. Proximal hypospadias
3. Penile curvature ≥30°
4. Syndromic anomalies or coagulopathy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Hypospadias Cosmetic Score (HOSE) | Follow-up evaluations will occur at 1, 3, and 6 months postoperatively.
  Assessment Method: Standardized digital photographs taken at 6 months postoperatively.
  Evaluators: Two independent pediatric urologists blinded to treatment allocation will evaluate the photographs.
  Measurement Tool: Cosmetic outcome scored using the Hypospadias Objective Scoring Evaluation (HOSE) system or a similar validated scale.
  Units: HOSE score (range 5-10).
  Higher scores: Indicate better cosmetic outcomes.

SECONDARY OUTCOMES:
Clinical examination for postoperative complications (fistula, stenosis, ) | during follow-up visits at 1, 3, and 6 months post-surgery.
  Assessment Method: Physical examination conducted by a trained clinician during follow-up visits at 1, 3, and 6 months post-surgery.
  Measurement Tools: Visual inspection and palpation for fistula or stenosis; documentation of findings in standardized case report forms.
  Units/Scoring: Presence or absence of complications (binary: yes/no).
  Interpretation: Higher occurrence indicates worse outcome.

OTHER OUTCOMES:
Body Mass Index (BMI) | Patients will be followed at 1, 3, and 6 months postoperatively for
  Measurement Method: Calculated by dividing weight in kilograms by height in meters squared (kg/m²).
  Calculation Details: BMI is obtained by measuring the child's weight using a calibrated scale and height using a stadiometer during the clinic visit. The BMI value is then calculated using the formula:
  BMI
  = weight (kg) height (m) 2 BMI= height (m) 2
  weight (kg)
  Units: kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Abbas, MD, PhD, Study Chair — Sidra Medicine
Locations (1):
- National Children's Medical Center, Tashkent, City, Uzbekistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abbas TO. Evaluation of penile curvature in patients with hypospadias; gaps in the current practice and future perspectives. J Pediatr Urol. 2022 Apr;18(2):151-159. doi: 10.1016/j.jpurol.2021.12.015. Epub 2021 Dec 31. PMID 35031224
- [Background] Abbas TO. An objective hypospadias classification system. J Pediatr Urol. 2022 Aug;18(4):481.e1-481.e8. doi: 10.1016/j.jpurol.2022.05.001. Epub 2022 May 11. PMID 35644790
- [Background] Elnashar AM, Albishbishy M, Sheir H, Elayyouti M, Elsherbiny M, Elzohiri M, Ghazaly Waly ME, Elsaied A. Comparative Study Between Autologous Platelet-rich Fibrin Membrane and Local Flaps as Intervening Layer in Management of Distal Hypospadias. J Pediatr Surg. 2025 Jan;60(1):161994. doi: 10.1016/j.jpedsurg.2024.161994. Epub 2024 Oct 11. PMID 39461004
- [Background] Guinot A, Arnaud A, Azzis O, Habonimana E, Jasienski S, Fremond B. Preliminary experience with the use of an autologous platelet-rich fibrin membrane for urethroplasty coverage in distal hypospadias surgery. J Pediatr Urol. 2014 Apr;10(2):300-5. doi: 10.1016/j.jpurol.2013.09.026. Epub 2013 Nov 13. PMID 24325905
- [Background] Moraschini V, Miron RJ, Mourao CFAB, Louro RS, Sculean A, da Fonseca LAM, Calasans Maia MD, Shibli JA. Antimicrobial effect of platelet-rich fibrin: A systematic review of in vitro evidence-based studies. Periodontol 2000. 2024 Feb;94(1):131-142. doi: 10.1111/prd.12529. Epub 2023 Sep 22. PMID 37740425
- [Background] Kajbafzadeh AM, Abolghasemi H, Eshghi P, Alizadeh F, Elmi A, Shafaattalab S, Dianat S, Amirizadeh N, Mohseni MJ. Single-donor fibrin sealant for repair of urethrocutaneous fistulae following multiple hypospadias and epispadias repairs. J Pediatr Urol. 2011 Aug;7(4):422-7. doi: 10.1016/j.jpurol.2010.06.004. Epub 2010 Jul 15. PMID 20634140
- [Background] Soyer T, Cakmak M, Aslan MK, Senyucel MF, Kisa U. Use of autologous platelet rich fibrin in urethracutaneous fistula repair: preliminary report. Int Wound J. 2013 Jun;10(3):345-7. doi: 10.1111/j.1742-481X.2012.00983.x. Epub 2012 May 9. PMID 22568526